CLINICAL TRIAL: NCT02680288
Title: Lorcaserin Effects on Cocaine Craving and Drug-Reinforced Behavior
Brief Title: Lorcaserin Intra Venous Cocaine Effects
Acronym: LIVE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Midwest Biomedical Research Foundation (Other)
Responsible Party: Principal Investigator, KENNETH GRASING, Staff Physician, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MIRB#0016
Record Dates: First submitted 2016-02-05; First posted 2016-02-11 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Cocaine Use Disorders
Keywords: Psychostimulant, Craving, Cocaine.
MeSH Terms: interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oral Placebo (Placebo Comparator): Oral inert treatment
  Interventions: Other: Oral Placebo
- Active Treatment, Low-Dose (Experimental): Lorcaserin 10 mg, single dose
  Interventions: Drug: Lorcaserin, 10 mg
- Active Treatment, High-Dose (Experimental): Lorcaserin 20 mg, single dose
  Interventions: Drug: Lorcaserin, 20 mg

INTERVENTIONS:
Drug: Lorcaserin, 10 mg — Oral type 2C serotonergic agonist, low-dose
  Other Names: Belviq
  Arms: Active Treatment, Low-Dose
Drug: Lorcaserin, 20 mg — Oral type 2C serotonergic agonist, high-dose
  Other Names: Belviq
  Arms: Active Treatment, High-Dose
Other: Oral Placebo — Oral inert treatment
  Arms: Oral Placebo

SUMMARY:
This is a randomized, cross-over, single-blind, placebo-controlled, single-center, multiple-panel evaluation of the potential for oral lorcaserin to modify cocaine self-administration in a laboratory setting. To prevent unauthorized drug use, study medications will be administered as participants are confined during overnight stays at the Medical Center. Non-treatment-seeking, regular cocaine users will receive oral treatment with single doses of placebo, lorcaserin 10 mg (Panel 1), or lorcaserin 20 mg (Panel 2). Afterwards, the subjective and reinforcing effects of intravenous cocaine will be measured in a laboratory setting.

DETAILED DESCRIPTION:
Background

Serotonin (5-HT) is one of three brain monoamines that are widely distributed in the brain and play important roles in affect and goal-directed behaviors. Limbic structures that underlie behavior motivated by palatable food and drugs of abuse receive dense projections from brainstem serotonergic nuclei. In rats, light and sound cues associated with access to cocaine strongly stimulate drug-seeking behavior. Agonists for the type 2C serotonergic receptor (5-HT₂cR) attenuate this responding.8 Drug taking (cocaine self-administration) is also attenuated at 5-HT₂cR agonist doses similar to those that decrease food-reinforced responding and cause reductions in locomotor activity.

Lorcaserin is a novel and selective agonist of the 5-HT₂cR recently approved by the FDA for weight loss therapy. It acts selectively at this receptor subtype with minimal activation of 5-HT₂ᴀR or 5-HT₂ᴃR receptors. Based on initial clinical studies leading to its approval, lorcaserin is well tolerated and probably does not cause cardiac valve disease or other serious side effects. Even so, given the potential for serious adverse events, the FDA has limited its use to patients who are either obese or overweight with a medical complication such as hypertension. Whether or not lorcaserin will become generally accepted as a long-term treatment for obesity will depend on the results of ongoing post-marketing studies of cardiovascular outcome data.

Rationale In preclinical studies, agonists for the 5-HT₂cR potently attenuate cocaine-seeking behavior. Lorcaserin is a recently approved selective 5-HT₂cR agonist with an acceptable safety profile in humans. No published studies have reported its effects on cocaine-induced craving or drug-reinforced responding in humans.

Specific Aims:

1. Evaluate whether lorcaserin treatment attenuates the positive subjective effects of cocaine and drug-reinforced behavior.
2. Determine whether active treatment modifies cocaine- or script- induced craving.

Methods This is a randomized, cross-over, double-blind, placebo-controlled, single-center, multiple-panel evaluation of the potential for oral lorcaserin to modify cocaine self-administration in a laboratory setting. Up to 32 non-treatment-seeking, regular cocaine users will receive treatment with single doses of oral placebo, lorcaserin 10 mg (Panel 1), or lorcaserin 20 mg (Panel 2). Script-guided imagery of autobiographical memories will be developed based on experiences related to cocaine use, anger, and a neutral event. Following treatment with lorcaserin, script-induced emotional states will be assayed. Sampling doses of cocaine (0.0, 0.23, and 0.46 mg/kg) will be administered, and participants will choose between self-administering additional intravenous doses or receiving monetary alternatives. Detailed measures of the negative and positive subjective effects of intravenous infusions will also be made. As noncontingent infusions of cocaine are administered, the pharmacokinetics of cocaine and lorcaserin will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Is non-treatment-seeking and has used cocaine regularly for at least six months.
2. Has used cocaine by a rapid route of administration (smoked or intravenous injection), at least three times per week, for three of the preceding six weeks.
3. Is male or female, between 21 and 50 years old.
4. Is able to verbalize understanding of the consent form, able to provide written informed consent, and verbalize willingness to complete study procedures.
5. Is agreeable to the study schedule and likely to complete all interventions and measures.
6. Has a medical history, physical exam, and screening laboratory results that demonstrate no contraindication to participation.

Exclusion Criteria:

1. Has a history of a medical adverse reaction to cocaine or other psycho stimulants, including loss of consciousness, chest pain, cardiac ischemia, or seizure.
2. Has any current Axis I psychiatric disorder other than drug abuse or dependence.
3. Meets DSM-IV-TR criteria for dependence on opiates, benzodiazepines, alcohol, or other sedative-hypnotics.
4. Has received opiate-substitution therapy within two months prior to enrollment.
5. Has a current or past history of seizure disorder other than febrile seizures, including alcohol- or psycho stimulant- related seizures, or family history of seizure disorder.
6. Has a diagnosis of adult asthma or chronic obstructive pulmonary disease.
7. Has had head trauma that resulted in neurological sequelae (e.g., loss of memory for greater than 5 minutes).
8. Has a history of valvular heart disease, congestive heart failure, syncope, bradycardia, or any other cardiac condition.
9. Has a condition that increases the risk of cocaine-induced hypertension or ischemic heart disease, such as hypertension, hypercholesterolemia, renal disease (serum creatinine > 1.4 mg/dl), diabetes (fasting glucose level ≥ 100 mg/dl).
10. Has a history of jaundice, hepatitis, or laboratory evidence of hepatic insufficiency (total bilirubin ≥ 2.0, serum albumin ≤ 3.5 gm./dl); or current abnormalities of liver function testing with serologic evidence of hepatitis (serology and coagulation will be evaluated in individuals with aspartate transaminase or Alaine aminotransferase > 40 IU/L).
11. History of priapism or conditions that would predispose to priapism (sickle cell anemia, multiple myeloma, leukemia, Peyronie's disease, or other anatomical deformation of the penis).
12. Currently being treated for erectile dysfunction.
13. Has an unstable medical condition, which, in the judgment of investigators, would make participation hazardous, such as AIDS or active TB.
14. If female, is pregnant or lactating (nursing), not practicing adequate methods of contraception, or planning to become pregnant within one month of conclusion of the study.
15. Has current suicidal ideation as assessed by the SCID interview.
16. Has clinically significant ECG abnormalities, including QTc interval prolongation > 450 milliseconds in men or 480 milliseconds in women.
17. Has donated blood or participated in another clinical trial within 4 weeks of enrollment.
18. In the opinion of investigators, is expected to fail to complete the study protocol due to probable incarceration or relocation from the clinic area.
19. Has had known or suspected hypersensitivity to Lorcaserin.
20. Is currently being treated with an adrenergic receptor antagonist ('beta blocker').
21. Is currently receiving Lorcaserin, potential CYP2D substrates, or medications associated with the serotonin syndrome or neuroleptic-malignant syndrome (see Tables 8 and 9).
22. Has a significant potential for violent behavior, as assessed by the Structured Assessment of Violence Risk in Youth (SAVRY).23

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-09 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Cocaine-Induced 'High' | Day 1 of Lorcaserin Treatment
  Visual analogue scale rating of 'high' after receiving cocaine

SECONDARY OUTCOMES:
Cocaine-Induced Craving | Day 1 of Lorcaserin treatment.
  Visual analogue scale rating of 'How much do you WANT to use cocaine' after receiving intravenous cocaine

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W Grasing, MD, Principal Investigator — Midwest Biomedical Research Foundation
Locations (1):
- Kansas City VA Medical Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burmeister JJ, Lungren EM, Kirschner KF, Neisewander JL. Differential roles of 5-HT receptor subtypes in cue and cocaine reinstatement of cocaine-seeking behavior in rats. Neuropsychopharmacology. 2004 Apr;29(4):660-8. doi: 10.1038/sj.npp.1300346. PMID 14627998
- [Background] Cunningham KA, Fox RG, Anastasio NC, Bubar MJ, Stutz SJ, Moeller FG, Gilbertson SR, Rosenzweig-Lipson S. Selective serotonin 5-HT(2C) receptor activation suppresses the reinforcing efficacy of cocaine and sucrose but differentially affects the incentive-salience value of cocaine- vs. sucrose-associated cues. Neuropharmacology. 2011 Sep;61(3):513-23. doi: 10.1016/j.neuropharm.2011.04.034. Epub 2011 May 11. PMID 21575646
- [Derived] Pirtle JL, Hickman MD, Boinpelly VC, Surineni K, Thakur HK, Grasing KW. The serotonin-2C agonist Lorcaserin delays intravenous choice and modifies the subjective and cardiovascular effects of cocaine: A randomized, controlled human laboratory study. Pharmacol Biochem Behav. 2019 May;180:52-59. doi: 10.1016/j.pbb.2019.02.010. Epub 2019 Feb 24. PMID 30811963